CLINICAL TRIAL: NCT01250366
Title: A Multi-center, Sequential-cohort, Placebo-controlled, 7-day Treatment Period Study of the Safety and Pharmacokinetics of Multiple Ascending Oral Doses of INX-08189 in Chronically-infected Genotype 1 HCV, Treatment-naïve Subjects
Brief Title: Study of the Safety & PK of INX-08189 in Chronically-infected HCV, Treatment-naïve Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: AI472-002; INH-189-002 (Other: INH-189-002)
Record Dates: First submitted 2010-11-22; First posted 2010-11-30 (Estimated); Last update posted 2012-07-12 (Estimated); Status verified 2012-07

CONDITIONS: HCV (Genotype 1)
Keywords: Safety and Pharmacokinetics
MeSH Terms: conditions — Hepatitis C | interventions — BMS-986094; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Arm 1: INX-08189 (9 mg) or Placebo (Experimental)
  Interventions: Drug: INX-08189; Drug: Placebo matching with INX-08189
- Arm 2: INX-08189 (25 mg) or Placebo (Experimental)
  Interventions: Drug: INX-08189; Drug: Placebo matching with INX-08189
- Arm 3: INX-08189 (50 mg + 9 mg) or Placebo (Experimental)
  Interventions: Drug: INX-08189; Drug: Placebo matching with INX-08189
- Arm 4: INX-08189 (50 mg) or Placebo (Experimental)
  Interventions: Drug: INX-08189; Drug: Placebo matching with INX-08189
- Arm 5: INX-08189 (9 mg) or Placebo + Ribavirin (Experimental)
  Interventions: Drug: INX-08189; Drug: Placebo matching with INX-08189; Drug: Ribavirin
- Arm 6: INX-08189 (25 mg) or Placebo + Ribavirin (Experimental)
  Interventions: Drug: INX-08189; Drug: Placebo matching with INX-08189; Drug: Ribavirin
- Arm 7: INX-08189 (100 mg) or Placebo (Experimental)
  Interventions: Drug: INX-08189; Drug: Placebo matching with INX-08189

INTERVENTIONS:
Drug: INX-08189 — Capsules, Oral, 9 mg, Once Daily, 7 Days
  Arms: Arm 1: INX-08189 (9 mg) or Placebo
Drug: INX-08189 — Capsule, Oral, 25 mg, Once Daily, 7 days
  Arms: Arm 2: INX-08189 (25 mg) or Placebo; Arm 6: INX-08189 (25 mg) or Placebo + Ribavirin
Drug: INX-08189 — Capsules, Oral, 50 mg, Single Dose, 1 day
  Arms: Arm 3: INX-08189 (50 mg + 9 mg) or Placebo
Drug: INX-08189 — Capsules, Oral, 9 mg, Once daily, 6 days
  Arms: Arm 3: INX-08189 (50 mg + 9 mg) or Placebo
Drug: INX-08189 — Capsules, Oral, 50 mg, Once daily, 7 days
  Arms: Arm 4: INX-08189 (50 mg) or Placebo
Drug: INX-08189 — Capsules, Oral, 9 mg, Once daily, 7 days
  Arms: Arm 5: INX-08189 (9 mg) or Placebo + Ribavirin
Drug: INX-08189 — Capsules, Oral, 100 mg, Once daily, 7 days
  Arms: Arm 7: INX-08189 (100 mg) or Placebo
Drug: Placebo matching with INX-08189 — Capsules, Oral, 0 mg, Once daily, 7 days
Drug: Ribavirin — Capsules, Oral, 1000 or 1200 mg daily (delivered in weight-adjusted am/pm divided dose), 7 days
  Arms: Arm 5: INX-08189 (9 mg) or Placebo + Ribavirin; Arm 6: INX-08189 (25 mg) or Placebo + Ribavirin

SUMMARY:
The purpose of this study is to determine the Safety and Pharmacokinetics of Multiple Ascending Oral Doses of INX-08189 in Chronically-infected Genotype 1 HCV, Treatment-naïve Subjects.

DETAILED DESCRIPTION:
This is a multi-center, sequential-cohort, double-blind, placebo-controlled, multiple ascending dose, 7-day treatment study in chronically-infected genotype 1 HCV, treatment-naïve subjects.

Primary Objectives include:

Safety

• to evaluate the safety of ascending oral doses of INX-08189 given once a day for seven (7) days in chronically-infected genotype 1 HCV, treatment-naïve subjects

Pharmacokinetic

• to characterize the pharmacokinetic (PK) profile of multiple ascending oral doses of INX-08189 in chronically-infected genotype 1 HCV, treatment-naïve subjects

Pharmacodynamic

• to evaluate the relationship between the metrics of the reduction from baseline in serum HCV RNA and PK parameters of INX-08189 and the metabolite INX-08032

Efficacy

• to measure the maximal reduction in plasma HCV RNA by ascending oral dose level of INX-08189 given once a day for seven (7) days in chronically-infected genotype 1 HCV, treatment-naïve subjects

ELIGIBILITY:
Inclusion Criteria:

At the screening visit (Visit 1), subjects will meet the following criteria:

1. Males & females, 18 - 65 years of age inclusive(BMI of at least 18kg/m2 not exceeding 36kg/m2);
2. Diagnosis of chronic HCV by 1 previous PCR result prior to screening, with a positive HCV viral load of at least 100,000IU/ml at screening measured by quantitative PCR;
3. HCV genotype 1 per central lab testing report;
4. HCV treatment-naïve (defined as no prior treatment with interferon, pegylated interferon, ribavirin, or any HCV direct acting anti-viral drugs);
5. Liver biopsy consistent with chronic HCV infection but non-cirrhotic as judged by a pathologist (Knodell < 3, Metavir <2, Ishak <4, or Batts & Ludwig <2) within the last 2 years & before Visit 2 (biopsy can be done within screening period);
6. Negative urine drug screen for drugs of abuse at screening and Study Day -1 (methadone use allowed);
7. Females will have a negative serum βHCG pregnancy test at screening & negative urine dipstick pregnancy test upon entry to clinical unit on Study Day -1;
8. Agreement by both females of childbearing potential & males(who have not been surgically sterilized) to practice an acceptable method of birth control. Surgical sterilization of either female or male partner must have occurred at least 6 month prior to first dose & females must be post-menopausal for 2 years to be considered of non-child-bearing potential. Acceptable contraceptive methods include 1 of the following: Oral & implantable hormonal contraceptives by female at least 3 months prior to the 1st dose of Study Drug, IUD in place at least 6 months prior to first dose, barrier methods either diaphragm or condom with spermicide. (Abstinence is not an acceptable method of birth control, subjects who indicate sexual inactivity must agree to utilize birth control in the event of sexual activity);
9. Willing & able to complete all study visits and procedures, & able to communicate with the investigator & other personnel;
10. Signed informed consent form (ICF) executed prior to protocol screening assessments

Exclusion Criteria:

At the screening visit subjects will not meet any of the following criteria:

1. Advanced liver disease, cirrhosis, or with signs of decompensated liver disease such as variceal bleeding, ascites, hepatic encephalopathy, active jaundice (total bilirubin > 2, or other evidence of decompensated liver disease;
2. Co-infection with HBV or HIV (positive test for HBsAg or anti-HIV Ab);
3. Acute cardiac ischemia, unstable heart disease or clinically symptomatic cardiac abnormalities apparent on ECG & PE, or a QTcB interval at Visit 1 of ≥ to 450ms by Bazette's correction, or personal or family history of Torsades de pointes;
4. Use of the following medications concurrently or within the 30 days prior to Screening associated with QT prolongation: macrolides, antiarrhythmic agents, azoles, fluoroquinolones, & tricyclic anti-depressants (methadone use allowed);
5. Use of immunosuppressive or immune-modulating agents (including corticosteroids & immunosuppressive agents) or presence of an immunologically-mediated autoimmune disease (other than asthma) or history of organ transplantation (inhaled steroids for asthma & topical steroid for minor skin conditions allowed);
6. Use of strong CYP3A4-inhibiting protease inhibitors (specifically atazanavir, indinavir, nelfinavir, saquinavir, & ritonavir), strong CYP3A4 inhibitors (specifically clarithromycin, itraconazole, ketoconazole, nefazodone, telithromycin), or strong CYP3A4 inducers (specifically rifampin, efavirenz, etravirine, phenobarbital, phenytoin, & carbamazepine);
7. Absolute NEUT count of <1800 cells/mm3 (or < 1500 cells/mm3 for African Americans), or platelet count <130,000 cells/mm3, or hemoglobin <11g/dl for women and <13g/dl for men;
8. A history of abnormal thyroid function not adequately controlled (defined as TSH levels < 0.8 x LLN or > 1.2 x the ULN);
9. Serum creatinine concentration > 1.5 times the upper limit of normal, or albumin < 3g/dl;
10. Presence or history of severe, or uncontrolled, or hospitalization-requiring psychiatric disease including severe depression, suicide attempts or any severity of psychosis;
11. Any malignancy within the last 5 years other than treated cervical carcinoma in situ or treated basal cell carcinoma with no more than 20% risk of recurrence within 2 years;
12. Alcohol abuse (investigator assessment) within the past 2 years or an alcohol use pattern that will interfere with the study conduct;
13. Drug abuse (investigator assessment)within the last 6 months with exception of methadone;
14. Current lactation or breastfeeding;
15. Major surgery within 30 days prior Visit 1;
16. Participation in another clinical trial of an investigational drug or device within 6 months prior to visit 1;
17. Donation of blood or plasma within 30 days prior to Visit 1

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2010-10; Primary Completion 2011-03 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Safety will be evaluated in an integrated way on the basis of the Adverse Event profiles, changes in laboratory values (serum chemistry, hematology and urinalysis), ECG data, and vital signs, viral resistance testing and results of Physical Exams. | periodically over 14 days
PK parameters following administration of INX-08189 will be determined using concentration data obtained via the assay of INX-08189 and INX-08032 in plasma, and the analysis of INX-08032 in urine | periodically over 14 days
The primary efficacy outcome is the maximum change from baseline in HCV RNA following 7 days of dosing. | 7 days

SECONDARY OUTCOMES:
Secondary efficacy outcome measures include the change in HCV RNA over time during the seven days of dosing and during the follow-up period thereafter. Additionally, viral load changes will be compared across the two genotypes 1a and 1b. | 14 days

CONTACTS AND LOCATIONS:
Locations (4):
- United States (3):
  - Los Angeles, California
  - Plymouth, Minnesota
  - San Antonio, Texas
- San Juan, Puerto Rico